CLINICAL TRIAL: NCT00477165
Title: Effect of Citalopram on Clinical Symptoms and Visceral Sensitivity in Patients With Irritable Bowel Syndrome
Brief Title: Citalopram in Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Uri Ladabaum, Principle Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H10539-18502
Record Dates: First submitted 2007-05-18; First posted 2007-05-22 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Antidepressant; IBS; Serotonin-reuptake inhibitor; SSRI; Visceral sensitivity; Barostat; Quality of life; Depression
MeSH Terms: conditions — Irritable Bowel Syndrome; Depression | interventions — Citalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Citalopram (Experimental): One 20mg capsule per day for 4 weeks, then 2 capsules per day (40mg) for 4 weeks
  Interventions: Drug: Citalopram
- Placebo (Placebo Comparator): Identical to citalopram 20mg capsule. One capsule per day for 4 weeks, then 2 capsules per day for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Citalopram — 20mg/day for 4 weeks, then 40 mg/day for 4 weeks
  Other Names: Celexa; Cipramil
  Arms: Citalopram
Drug: Placebo — Identical to citalopram 20mg capsules; 1 capsule/day for 4 weeks, then 2 capsules/day for 4 weeks
  Arms: Placebo

SUMMARY:
Hypotheses:

1. Primary null hypothesis: The rate of clinical response, assessed as patient-reported global symptom rating and "adequate relief of IBS symptoms," does not differ between non-depressed IBS patients treated with the SSRI citalopram and patients treated with placebo.
2. Secondary null hypotheses:

   1. Changes in disease-related quality of life, assessed with the IBS-QOL instrument, do not differ between patients treated with the SSRI citalopram and patients treated with placebo.
   2. Changes in rectosigmoid visceral sensitivity, assessed by barostat balloon distention, do not differ between patients treated with the SSRI citalopram and patients treated with placebo.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) affects an estimated 15 million Americans at a cost of $1.7 billion per year. Visceral hypersensitivity is present in many patients with IBS, but its contribution to clinical symptoms is unclear. Tricyclic antidepressants may be beneficial in IBS, but their side effects can be unacceptable. Because they are better tolerated, selective serotonin reuptake inhibitors (SSRIs) are often used to treat IBS, but their efficacy in IBS has not been examined in controlled studies. We propose a randomized, placebo-controlled trial of SSRI treatment in IBS. Non-depressed patients will be studied in order to assess SSRI effects on IBS independent of depression. Our specific aims are: 1) To determine whether the SSRI citalopram is superior to placebo in improving clinical symptoms, disease-related quality of life, and tolerance to rectal balloon distension; 2) To assess whether symptomatic improvement is correlated with improvement in quality of life and/or visceral sensitivity. Subjects will fulfill Rome II IBS criteria, will have normal screening studies, and will not be depressed or on antidepressants. Global and specific symptoms, and satisfaction will be rated daily during a 1-week baseline. Subjects will then be randomized in concealed, double-blind fashion to citalopram or placebo, will complete the validated IBS-QOL instrument, and will undergo rectal compliance and sensory testing with a barostat. Subjects will be treated and will rate symptoms and satisfaction weekly for a total of 8 weeks, and also daily during the final week for comparison with the baseline. At study end, subjects will again complete the IBS-QOL and undergo a barostat study. For the primary outcome, we estimate that to detect a standardized effect size of 0.9 in global symptom rating with 2-sided α=0.05 and β=0.1, 54 subjects are needed. We plan to enroll 60 subjects, which will allow detection of an odds ratio for response (adequate relief) of 4.5 with 2-sided α=0.05 and β=0.2. If the odds ratio for this dichotomous outcome is smaller, this study will provide pilot data for a larger trial. Clinical symptoms are expected to fluctuate. Even if citalopram is not superior to placebo, prospectively collected data will illuminate the relationship between symptoms and visceral sensitivity, and the placebo effect.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria are:

1. Fulfilling Rome II IBS definition;
2. Age ≥18 yrs and able to give informed consent;
3. Normal sigmoidoscopy, colonoscopy or barium enema within 5 years, normal complete blood count and thyroid studies, and negative stool ova and parasite exam for patients with diarrhea.

Exclusion Criteria:

Exclusion criteria are:

1. Current psychiatric diagnosis or active treatment with antidepressants;
2. Pregnancy;
3. Major systemic illness, or illness that could explain IBS-like symptoms;
4. Active IBS therapy other than fiber or loperamide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2001-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uri Ladabaum, M.D., M.S., Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 234 potentially eligible subjects were identified. Of these, 180 were excluded and 54 enrolled in the study, with 27 each randomized to citalopram and placebo.
Groups:
- Cialopram: One 20mg capsule per day for 4 weeks, then 2 capsules per day (40mg) for 4 weeks
Period: Overall Study
Arm/Group | Cialopram | Placebo
Started | 27 | 27
Completed | 20 | 25
Not Completed | 7 | 2
Not completed — Adverse Event | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cialopram | Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Continuous [Mean (Full Range); unit: years] | 53 [27 to 75] | 51 [30 to 75] | 52 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Who Self-reported "Adequate Relief"
Description: Participants were asked weekly to answer subjectively whether weekly adequate relief from IBS symptoms was achieved. Overall response was defined as having achieved adequate relief in at least 3 of the past 6 weeks.
Time Frame: Baseline, weekly for 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 27 | 27
Participants | 12 | 15
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Null hypothesis: number of patients achieving adequate relief is the same in both Citalopram and Placebo groups; Test type: Superiority or Other; p = 0.59, t-test, 2 sided — p<0.05 for statistical significance; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.687 to 1.196] — Repeated-measures logistic regression model, assuming the citalopram effect builds linearly over time starting at week 3

2. Secondary Outcome: Change From Baseline in IBS-QOL Score at Week 8
Description: The IBS-QOL is a self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. The IBS-QOL consists of 34 statements about bowel problems, each with a five-point response scale ranging from 1 (no problems) to 5 (most problems). The individual scores are summed and averaged for a total score, then transformed to a 0-100 scale for ease of interpretation with higher scores indicating better IBS-specific quality of life.
Time Frame: Baseline; Week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 27 | 27
units on a scale | 6.3 [-0.07 to 12.7] | 7.6 [2.4 to 12.9]

3. Secondary Outcome: Mean Sensation Score as a Function of Distending Pressure at the End of the Study
Description: A 500mL polyethylene bag was passed into the rectum, with tubing connected to a barostat, which was controlled by a computer that recorded bag pressure, volume, and corrected volume every second. After 5 minutes, the bag was unfurled with 100mL of air and deflated; with inflations lasting 45 seconds from 0 up to 60 mmHg, increasing by 3 mmHg, and separated by 45-second deflations, subjects rated sensation 30 seconds into each inflation. Sensation score scale: 0=no inflation sensation, 1-5=increasing painless sensation, 6=threshold pain, 10=worst imaginable pain.
Time Frame: Week 8
Population: Participants with available data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 20 | 25
units on a scale
  Distending pressure 12mmHg | 1 [1 to 2] | 2 [2 to 3]
  Distending pressure 24mmHg | 4 [3 to 5] | 6 [3 to 6]
  Distending pressure 36mmHg | 5 [4 to 7] | 7 [5 to 9]
  Distending pressure 48mmHg | 7 [5 to 8] | 6 [4 to 10]

4. Secondary Outcome: Urgency Score as a Function of Distending Pressure at the End of the Study
Description: A 500mL polyethylene bag was passed into the rectum, with tubing connected to a barostat, which was controlled by a computer that recorded bag pressure, volume, and corrected volume every second. After 5 minutes, the bag was unfurled with 100mL of air and deflated; with inflations lasting 45 seconds from 0 up to 60 mmHg, increasing by 3 mmHg, and separated by 45-second deflations, subjects rated urgency for bowel movement 30 seconds into each inflation. Urgency score scale: 0=no urgency, 1=threshold urgency, 5=worst imaginable urgency.
Time Frame: Week 8
Population: Participants with available data were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 20 | 25
units on a scale
  Distending pressure 12mmHg | 1 [1 to 2] | 2 [1 to 2]
  Distending pressure 24mmHg | 4 [3 to 4] | 5 [4 to 5]
  Distending pressure 36mmHg | 4 [4 to 5] | 5 [4 to 5]
  Distending pressure 48mmHg | 5 [4 to 5] | 5 [4 to 5]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: During the study, subjects were asked to call a research coordinator weekly to report completion of questionnaires. If the telephone call was not received, a research coordinator contacted the subject. Subjects were asked to call if they experienced side effects.
Arm/Group | Citalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 7/27 | 2/27
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=27) | Placebo (N=27)
Fatigue (General disorders) | 3 (3) | 0 (0) — decreased energy
Insomnia (General disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Somnolence (Psychiatric disorders) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — pregnancy despite birth control

LIMITATIONS AND CAVEATS:
Results have been entered as available in the published manuscript; the PI is no longer at UCSF. This trial has the limitation of relatively small sample size. A potential limitation is that patients could have been unblinded based on side effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes